CLINICAL TRIAL: NCT00683319
Title: CCLG Observational Study of the Outcome of Ependymoma in Infants Diagnosed Before Their Third Birthday
Brief Title: Observing Young Patients With Ependymoma Undergoing Standard Combination Chemotherapy
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000590666; CCLG-CNS-2007-09; EU-20835
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2009-06

CONDITIONS: Brain and Central Nervous System Tumors; Cognitive/Functional Effects; Long-term Effects Secondary to Cancer Therapy in Children; Ototoxicity
Keywords: long-term effects secondary to cancer therapy in children; cognitive/functional effects; ototoxicity; childhood infratentorial ependymoma; childhood supratentorial ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Ototoxicity | interventions — Carboplatin; Cisplatin; Cyclophosphamide; Methotrexate; Vincristine; Chemotherapy, Adjuvant; Mental Status and Dementia Tests; Magnetic Resonance Spectroscopy

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: methotrexate
Drug: vincristine sulfate
Procedure: adjuvant therapy
Procedure: cognitive assessment
Procedure: magnetic resonance imaging
Procedure: magnetic resonance spectroscopic imaging
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Gathering information about how young patients with ependymoma respond to standard combination chemotherapy and learning about the long-term effects of this treatment may help doctors plan better treatment.

PURPOSE: This phase III trial is observing young patients with ependymoma undergoing standard combination chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the overall survival and event-free survival of all infants diagnosed with ependymoma before their third birthday.
* To determine the overall survival and event-free survival of infants diagnosed with ependymoma before their third birthday when treated with standard chemotherapy comprising vincristine, carboplatin, high-dose methotrexate, cyclophosphamide, and cisplatin.

Secondary

* To investigate the reasons why the primary tumor was completely resected in patients who were able to undergo complete resection of the tumor.
* To continue to investigate the biological characteristics of ependymoma.
* To correlate functional imaging studies of ependymoma with biological characteristics of the tumor.
* To provide a standard treatment regimen for patients with residual disease after optimal surgery who have already participated in a phase II study.
* To prospectively document renal function, hearing, and neurocognitive late effects after completion of study treatment.

OUTLINE: This is a multicenter study. Patients are stratified according to extent of prior surgical resection and presence of metastatic disease (complete resection of tumor vs metastatic disease at diagnosis vs no complete resection of tumor).

Patients receive vincristine IV on days 1, 15, and 29, carboplatin IV over 1 hour on day 1, high-dose methotrexate* IV over 24 hours on day 15, cyclophosphamide IV over 1 hour on day 29, and cisplatin IV over 48 hours on days 43 and 44. Treatment repeats every 8 weeks for 7 courses in the absence of disease progression or unacceptable toxicity. Patients with residual disease after completion of treatment may receive other treatment at the discretion of the investigator.

NOTE: *Patients initially treated on clinical trial CCLG-CNS-2005-03 who have no residual disease do not receive high-dose methotrexate in courses 5-7.

Patients undergo observational assessments comprising physical and neurological examination; MRI/ MRS scanning of the head and spine; and audiology, renal, endocrine, neurocognitive, and quality of life evaluations periodically for at least 5 years after the completion of study treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed WHO grade 3 anaplastic (malignant) ependymoma or WHO grade 2 ependymoma, including the following variants:

  * Papillary
  * Cellular
  * Clear cell
  * Tanycytic
* No myxopapillary ependymoma, subependymoma, or ependymoblastoma
* Meets 1 of the following criteria:

  * Has undergone complete resection of the primary tumor (prior to starting chemotherapy)

    * Two or more surgical procedures to achieve complete resection allowed
  * Metastatic disease at diagnosis (with or without complete resection of the primary tumor)
  * Unable to undergo complete resection of the primary tumor (with or without metastatic disease)
* Patients with measurable residual disease (primary or metastatic disease) are eligible provided they undergo treatment on clinical trial CCLG-CNS-2005-03 prior to entering this study
* Has undergone surgical resection OR completed treatment on clinical trial CCLG-CNS-2005-03 within the past 3 weeks
* Patients who are unable to tolerate chemotherapy or who do not receive treatment according to the CCLG guidelines for ependymoma due to parental preference or recommendation from the treating physician are eligible

PATIENT CHARACTERISTICS:

* Able to tolerate IV hydration
* No active infection

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2008-04; Primary Completion 2034-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival
Event-free survival
Response to chemotherapy, if there is residual disease
Requirement for radiotherapy (i.e., residual disease at the completion of chemotherapy, progressive disease during chemotherapy, or recurrent disease during or after completion chemotherapy)
Late effects of treatment (i.e., ototoxicity and nephrotoxicity at the completion of chemotherapy and neurocognitive outcomes at 5, 7, 11, and 16 years of age)

CONTACTS AND LOCATIONS:
Overall Officials: Martin W. English, MD, Principal Investigator — Birmingham Children's Hospital
Locations (10):
- United Kingdom (10):
  - Birmingham Children's Hospital, Birmingham, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Queen's Medical Centre, Nottingham, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland